CLINICAL TRIAL: NCT01529294
Title: Open-label, Single-dose, Parallel-group Study to Compare the PKs of Iloperidone in Subjects With Mild or Moderate Hepatic Impairment With That in Matched Healthy Control Subjects
Brief Title: Single-dose Iloperidone Pharmacokinetics in Patients With Mild or Moderate Liver Disease, Compared to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: CILO522D2401
Record Dates: First submitted 2011-09-23; First posted 2012-02-08 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment; Iloperidone; ILO522D; Pharmacokinetics
MeSH Terms: interventions — iloperidone

ARMS (1):
- Iloperidone (Experimental): Eligible subjects receive a single oral dose of 2 mg iloperidone as a tablet
  Interventions: Drug: Iloperidone

INTERVENTIONS:
Drug: Iloperidone

SUMMARY:
This study aims to determine the pharmacokinetic profile and the tolerability of iloperidone in subjects with mild or moderate hepatic impairment comparatively to healthy matched subjects

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (all subjects):
* Caucasian subjects
* Inclusion criteria (hepatic impaired subjects):
* subjects with physical signs consistent with a clinical diagnosis of stable liver disease, which has been confirmed by imaging techniques, ultrasound, Magnetic Resonance Imaging or Computed Tomogram within 3 months of screening, and a creatinine clearance > 50 mL/min (based on Cockroft and Gault formula).
* Inclusion criteria (healthy volunteers):
* good general health
* matched by age, gender, smoking status, Body Mass Index, and CYP2D6 phenotype to hepatic impaired subjects.

Exclusion Criteria:

* Exclusion criteria (all subjects):
* Subjects who report smoking a pipe, cigars or more than 20 cigarettes per day .
* History of drug abuse as defined in Diagnostic and Statistical Manual of Mental Disorders, Diagnostic Criteria for Drug and Alcohol Abuse, within the 12 months prior to screening
* History of first-dose response/syncope to alpha1-blocking agents
* Exclusion criteria (Hepatic impaired subjects):
* Patients with symptoms or 6 months past history of encephalopathy.
* Patients with clinical evidence of moderate-severe ascites.
* Patients having a previous surgical porto-systemic shunt.
* Exclusion criteria (Healthy volunteers):
* History of alcohol abuse prior to dosing, or evidence of such abuse during screening.
* Pulse Rate > 200 msec

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Measure: Area Under Curve (AUClast, AUCinf) and maximum concentration (Cmax) | predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96 and 120 hours post-dose
  Pharmacokinetics of iloperidone in subjects with mild or moderate hepatic impairment, compared to healthy volunteers.
Maximum plasma concentration following drug administration (Cmax) of iloperidone | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose, and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentration will be measured.
Protein binding of iloperidone | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose, and from pre-dose to 48 hours post-dose
  Blood samples will be collected and protein binding will be measured .
Area under the plasma concentration-time Curve from time zero to infinity (AUCinf) of iloperidone | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose, and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentration will be measured.

SECONDARY OUTCOMES:
Area Under the plasma Curve (AUC) of iloperidone metabolite P88 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentrations of metabolite 88 will be measured
Area under the plasma concentration-time Curve from time zero to infinity (AUCinf) of iloperidone metabolite P88 records, listed by subject. Summary statistics provided by impairment group and visit/time. | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentrations of metabolite 88 will be measured
Maximum plasma concentration following drug administration (Cmax) of iloperidone metabolites P88 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentrations of metabolite 88 will be measured
Protein binding of iloperidone metabolites P88 (CLr) | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood samples will be collected and protein binding of metabolite 88 will be measured
Area Under the plasma Curve (AUC) of iloperidone metabolite P95 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentrations of metabolite 95 will be measured
Area under the plasma concentration-time Curve from time zero to infinity (AUCinf) of iloperidone metabolite P95 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentrations of metabolite 95 will be measured
Maximum plasma concentration following drug administration (Cmax) of iloperidone metabolites P95 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood and urine samples will be collected and plasma and urine concentrations of metabolite 95 will be measured
Protein binding of iloperidone metabolites P95 | pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 hours post-dose and from pre-dose to 48 hours post-dose
  Blood samples will be collected and protein binding of metabolite 95 will be measured
Number of participants with adverse events | Day 6
  Adverse events will be determined by evaluating clinical, laboratory evaluations, impact on vital signs and impacts on Electrocardiograms (ECGs)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- United States (4):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, South Miami, Florida